CLINICAL TRIAL: NCT04888455
Title: The Influence of Sensory Phenotype on the Risk of Developing Neuropathic Pain
Brief Title: DOLORisk: Research on Risk Factors and Determinants for Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: University of Kiel (Other)
Collaborators: Horizon 2020 - European Commission (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Oxford (Other); Imperial College London (Other); Technion, Israel Institute of Technology (Other); University of Aarhus (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Janne Gierthmuhlen, Prof. Dr. med., University of Kiel
Other Study IDs: 633491 - DOLORisk WP4
Record Dates: First submitted 2021-05-05; First posted 2021-05-17 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Neuropathic Pain
Keywords: pain prevention; painful neuropathy,; painless neuropathy; QST; patient-reported outcomes; PRO
MeSH Terms: conditions — Neuralgia; Neuropathy, Painful

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Painful neuropathy: Patients with presence of probable (presence of a combination of symptoms and signs of neuropathy include any two or more of the following: neuropathic symptoms, decreased distal sensation, or unequivocally decreased or absent ankle reflexes) or confirmed (presence of an abnormality of NC or validated measure of small fiber neuropathy with class 1 evidence with corresponding symptoms) neuropathy AND with probable or definite neuropathic pain according to the NeuPSIG algorithm.
  Interventions: Diagnostic Test: Quantitative sensory testing (QST)
- Painless neuropathy: Patients with presence of probable (presence of a combination of symptoms and signs of neuropathy include any two or more of the following: neuropathic symptoms, decreased distal sensation, or unequivocally decreased or absent ankle reflexes) or confirmed (presence of an abnormality of NC or validated measure of small fiber neuropathy with class 1 evidence with corresponding symptoms) neuropathy AND with unlikely neuropathic pain according to the NeuPSIG algorithm.
  Interventions: Diagnostic Test: Quantitative sensory testing (QST)

INTERVENTIONS:
Diagnostic Test: Quantitative sensory testing (QST) — Demographic data, pain characteristics, health status, emotional well-being, personality and lifestyle are assessed by questionnaires. Additionally, all patients underwent a clinical neurological examination and quantitative sensory testing (QST) according to the German Research Network on Neuropathic Pain (DFNS).
  Other Names: Different Questionnaires

SUMMARY:
Patients with neuropathic pain of multiple etiologies and a control cohort of patients with the same neuropathic entities who did not develop neuropathic pain are examined clinically, phenotyped with QST and questionnaires. Both groups are analyzed in order to find risk factors for painful neuropathy.

DETAILED DESCRIPTION:
Patients with probable (presence of a combination of symptoms and signs of neuropathy include any two or more of the following: neuropathic symptoms, decreased distal sensation, or unequivocally decreased or absent ankle reflexes) or confirmed (presence of an abnormality of NC or validated measure of small fiber neuropathy with class 1 evidence with corresponding symptoms) neuropathy are included. Patients are then further divided into those with painful and painless neuropathy according to the NeuPSIG algorithm. Patients with probable or definite neuropathic pain are classified as painful neuropathy, those with unlikely neuropathic pain classified as painless neuropathy (with concomitant nociceptive pain of other origin, e.g. headache etc.). Patients with possible neuropathic pain are excluded from analysis as are patients with skin lesions or dermatological disorders in the areas to be tested upon QST, with any painful or neurological comorbidity that could otherwise influence testing results such as vascular disease, radiculopathy, spinal canal stenosis etc. Inclusion was restricted to patients with polyneuropathy to make the investigated patient sample as homogenous as possible.

Age, gender, BMI, ethnicity, years in education, family history of chronic pain, etiology of neuropathy, presence of early traumatic events and hospital admissions, smoking and alcohol habits, pain characteristics (von Korff, BPSI, NPSI), emotional well-being (PROMIS depression/ anxiety), personality (TIPI, IPIP, PCS), severity of neuropathy are assessed and QST performed.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of Polyneuropathy

Exclusion Criteria:

* Patients with polyneuropathy and possible neuropathic pain
* Patients with skin lesions or dermatological disorders in the areas to be tested upon QST
* Patients with any painful or neurological comorbidity that could otherwise influence testing results such as vascular disease, radiculopathy, spinal canal stenosis etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In- and outpatients with presence of probable (presence of a combination of symptoms and signs of neuropathy include any two or more of the following: neuropathic symptoms, decreased distal sensation, or unequivocally decreased or absent ankle reflexes) or confirmed (presence of an abnormality of NC or validated measure of small fiber neuropathy with class 1 evidence with corresponding symptoms) neuropathy. Patients are then further divided into those with painful and painless neuropathy according to the NeuPSIG algorithm.
Sampling Method: Probability Sample
Enrollment: 1550 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Presence of Pain measured by Pain severity | through study completion, an average of 2 years
  Measurement on NRS [NRS 0-10]

SECONDARY OUTCOMES:
Severity of Neuropathy measured by Toronto Neuropathy scale | through study completion, an average of 2 years
  Total Score [0-19 points] from history and clinical examination
Somatosensory phenotype measured by Quantitative sensory testing | through study completion, an average of 2 years
  Assessment of somatosensory phenotype with the protocol of the German REsearch Network of Neuropathic Pain (DFNS)
Emotional well-being | through study completion, an average of 2 years
  assessed by anxiety PROMIS Short Form v1.0 -Anxiety 6a, Depression 6a, Fatigue and Sleep
Personality characteristics | through study completion, an average of 2 years
  assessed by Ten-Item Personality Inventory and International Personality Item Pool's
Pain Catastrophizing | through study completion, an average of 2 years
  assessed by Pain Catastrophizing scale (PCS) total score [0-52 points]
Presence of family history of chronic pain | through study completion, an average of 2 years
  Presence of pain in family

CONTACTS AND LOCATIONS:
Overall Officials: David Bennett, Prof., Study Director — University of Oxford
Locations (1):
- University of Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pascal MMV, Themistocleous AC, Baron R, Binder A, Bouhassira D, Crombez G, Finnerup NB, Gierthmuhlen J, Granovsky Y, Groop L, Hebert HL, Jensen TS, Johnsen K, McCarthy MI, Meng W, Palmer CNA, Rice ASC, Serra J, Sola R, Yarnitsky D, Smith BH, Attal N, Bennett DLH. DOLORisk: study protocol for a multi-centre observational study to understand the risk factors and determinants of neuropathic pain. Wellcome Open Res. 2019 Feb 1;3:63. doi: 10.12688/wellcomeopenres.14576.2. eCollection 2018. PMID 30756091
- [Derived] Gierthmuhlen J, Attal N, Baskozos G, Bennedsgaard K, Bennett DL, Bouhassira D, Crombez G, Finnerup NB, Granovsky Y, Jensen TS, John J, Kennes LN, Laycock H, Pascal MMV, Rice ASC, Shafran-Topaz L, Themistocleous AC, Yarnitsky D, Baron R. What is associated with painful polyneuropathy? A cross-sectional analysis of symptoms and signs in patients with painful and painless polyneuropathy. Pain. 2024 Dec 1;165(12):2888-2899. doi: 10.1097/j.pain.0000000000003310. Epub 2024 Jul 3. PMID 38968400
- See also: Study protocol — https://pubmed.ncbi.nlm.nih.gov/30756091/